CLINICAL TRIAL: NCT00301171
Title: Respiratory Function in Infants With Persistent Wheezing
Brief Title: Treatment of Persistent Wheezing in Infants and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 370; K23HL067881-04 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2007-12

CONDITIONS: Asthma; Respiratory Sounds
Keywords: Wheezing
MeSH Terms: conditions — Asthma; Respiratory Sounds

INTERVENTIONS:
Drug: Inhaled Fluticasone

SUMMARY:
Wheezing is a high-pitched whistling sound that is produced when air flows through narrowed lung airways. It is a common symptom of asthma. Persistent wheezing is commonly treated with bronchodilators and inhaled steroids; however, when wheezing is temporarily caused by a virus or exposure to tobacco smoke, this may not be the most effective treatment. The purpose of this study is to evaluate the cause of wheezing in infants and children and to assess the effectiveness of inhaled steroids on improving lung function.

DETAILED DESCRIPTION:
Asthma prevalence has steadily increased in the United States since the early 1980s, with infants and young children showing the largest increase. Some young children experience wheezing, but it is not known if this is related specifically to asthma. Wheezing may be caused by a respiratory syncytial virus, maternal smoking, a family history of asthma, or allergies. In addition, some infants who experience wheezing may have small or dysfunctional airways and may not respond well to commonly prescribed anti-inflammatory medications. Because of the many causes of wheezing, in order to prescribe the most effective treatment, it is necessary to thoroughly assess lung function, allergic sensitization, and airway inflammation. The purpose of this study is to examine the causes of moderate to severe wheezing in infants and assess the infants' response to inhaled corticosteroid therapy. The study will also assess new and safer ways to measure lung function and airway inflammation.

This study will enroll infants with moderate to severe persistent wheezing. At study entry, participants will undergo lung function testing, which will include a spirometry test, measures of lung volumes, and assessment of bronchodilator responsiveness. Exhaled breath condensate and blood will be collected, and skin-prick testing will be performed to test for allergies. Participants will then be randomly assigned to receive either fluticasone, an inhaled steroid, or placebo for one month. At the end of the month, lung function testing will be performed and exhaled breath and serum measures will be collected to assess airway inflammation. Participants will attend a follow-up evaluation at age 5 years. During the evaluation, lung function, exhaled breath condensate, and serum markers of inflammation will be measured again, and skin-prick testing will also be performed again.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe persistent wheezing, as defined by the National Asthma Education and Prevention Program Expert Panel Report 2
* No signs of upper or lower respiratory tract infection for at least two weeks prior to study entry

Exclusion Criteria:

* Received therapy with inhaled corticosteroids in the month prior to study entry
* History of seizures or other neurologic disorders
* Hypoxemia requiring supplemental oxygen to maintain oxygen saturation above 90%
* Sepsis
* Underwent a tracheostomy
* Heart disease
* Suspected or documented pulmonary hypertension
* Currently undergoing assisted ventilation
* Born at less than 36 weeks gestation

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2003-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in FEF75 levels
Change in RV/TLC ratio
Loss of bronchodilator responsiveness (measured at the end of the one month treatment period and follow-up evaluation when participant is 5 years of age)

SECONDARY OUTCOMES:
Change in asthma symptom scores (measured at the end of the one month treatment period and follow-up evaluation when participant is 5 years of age)

CONTACTS AND LOCATIONS:
Overall Officials: Amy G. Filbrun, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States